CLINICAL TRIAL: NCT04312646
Title: Added Value of Ultrasound Elasatography in Characterization of Thyroid Nodules
Brief Title: Elastography in Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omima mahran hussein abd el wadod, principal investigator, Assiut University
Other Study IDs: ultrasound in thyroid nodules
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with thyroid nodules
  Interventions: Device: Elastography .

INTERVENTIONS:
Device: Elastography . — Performance of US, elastography

SUMMARY:
Thyroid nodules are a common finding in the general population,however, they are mostly unpalpable and usually discovered either during neck ultrasound (US) examination or by pathological examination at autopsy. They are found in about 8% of adults. Most thyroid nodules ''incidentalomas" are benign, however 7% may be malignant. Early detection of thyroid cancer helps in early treatment and better survival US is an accurate method for detection of thyroid nodules; however, US has a low accuracy in differentiating between benign from malignant thyroid nodules . US could suggest a malignancy likelihood criteria of a thyroid nodule, such as hypoechogenicity, increased intranodular vascularity, irregular margins, microcalcifications, absent halo, and a taller-than-wide shape measured in the transverse dimension.

DETAILED DESCRIPTION:
US elastography has been used to detect the nature of thyroid nodules, by measuring the tissue stiffness non invasively. It depends on tissue deformation strain that is caused by external compression.it is complementary to gray scale findings particularly in nodules with indeterminate US findings, also US elastography could be used to guide the follow up of leisons diagnosed as benign at ( FNA) fine needle aspiration .

There are two main thyroid elastography methods in clinical practice: strain elastography (SE) and shear-wave elastography (SWE) .

Elastography methods can be classified into different variants based on the excitation method (external force, internal force, and acoustic radiation force [ARF]), and how stiffness is expressed . (A) strain elastography . SE reqires mechanical stress, which results in axial displacement of the tissue Tissue deformation from the stress is measured and visualized on a screen. The main limitations of SE are operator dependence for the angle, strength, and duration of compression.

(B) shear wave elastography . The acoustic pulses from the probe stimulate the target tissue, creating a shear wave (SW) traveling perpendicular to the conventional US waves. SWs are the transverse components of particle displacement that are rapidly attenuated by the tissue (1- 10 m/sec). This transverse component is tracked and measured as a numerical value corresponding to the shear-wave speed (SWS).This speed is closely related to the Young modulus formula, in which tissue elasticity can be assessed from the SW propagation.

US elastography is completely painless for the patient, and only requires a few extra minutes, with no separate patient preparation. US elastography has the potential to distinguish benign from malignant TNs, offering non-invasive complementary information to conventional US.

It may be particularly useful in patients who have nondiagnostic or indeterminate FNA cytology results.

ELIGIBILITY:
Inclusion Criteria:

* solitary nodule on clinical or ultrasound examination

Exclusion Criteria:

* Patients received any medical treatment or chemo or radiotherapy.
* Patients underwent fine needle aspiration cytology or biopsy
* Nodules with calcification and cystic changes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with solitary thyroid nodule
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of Elastography in differentiation between benign and malignant thyroid nodules | one year
  by its additional information over the classic gray scale and color Doppler ultrasound

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787